CLINICAL TRIAL: NCT05227014
Title: Enhanced Recovery and Patient Blood Management in Colorectal Surgery: the Italian ColoRectal Anastomotic Leakage Study Group (iCral 4).
Brief Title: Enhanced Recovery and Patient Blood Management in Colorectal Surgery
Acronym: iCral4
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Sandro Pertini, Roma (Other)
Collaborators: Associazione Chirurghi Ospedalieri Italiani (Other)
Responsible Party: Principal Investigator, Marco Catarci, Director, General Surgery Unit, Ospedale Sandro Pertini, Roma
Other Study IDs: iCral4
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Anastomotic Leak; Colorectal Neoplasms; Blood Transfusion Complication; Colorectal Disorders
Keywords: PBM; ERAS
MeSH Terms: conditions — Anastomotic Leak; Colorectal Neoplasms; Transfusion Reaction | interventions — Colectomy; Proctectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colorectal resection — All patients undergoing elective colorectal surgery with anastomosis will be included in a prospective database after written informed consent.
  Other Names: Colectomy, proctectomy

SUMMARY:
To prospectively study the effect of adherence to ERAS and PBM programs on early outcomes after colorectal surgery

DETAILED DESCRIPTION:
The ultimate goal of any surgery is to return the patient to his baseline functional status, if not an improved one, as rapidly as possible and with the least amount of intercurrent disability. Enhanced Recovery After Surgery (ERAS) is a multimodal and multifactorial approach to the optimization of perioperative management. In order to modify and improve the response to surgery-induced trauma, the program relies on a series of evidence-based items related to pre-, intra- and post-operative care. Preoperative anemia is a contraindication to elective surgery. Nonetheless, it is very common, affecting up to 39% of patients candidate to general surgery. Logically, it is the strongest predictor of blood transfusions (five-fold) in the post-operative period and it is associated to several risks and significant morbidity, such as infections (two-fold) and kidney injury (four-fold), as well as a 22% longer hospital stay. More importantly, peri-operative anemia is now recognized as strongly and independently related to post-operative mortality (adjusted odd ratio 2.36), also besides blood transfusions. Post-operative anemia regards up to 90% of patients after major surgery. The immediate and most widely used treatment for post-operative anemia is blood transfusion. Blood transfusions carry several complications, culminating in a high incidence of morbidity and mortality. In particular, they are related to increased length of hospital stay and rate of discharge to an inpatient facility, worse surgical and medical outcomes, allergic reactions, transfusion-related acute lung injury, volemic overload, venous thromboembolism, graft versus host disease, immunosuppression, and post-operative infections. Two previous prospective studies of the Italian ColoRectal Anastomotic Leakage (iCral) study group identified intra- and post-operative blood transfusions as an independent factor with negative influence on all early outcomes after colorectal surgery. In particular, they resulted as a major independent determinant of anastomotic leakage.

In recent years, various strategies have been studied to reduce the use of blood transfusions to prevent transfusion-related adverse events, increase patient safety, and reduce costs. As a consequence, a new concept was born: the patient blood management (PBM). According to the World Health Organization (WHO), PBM is defined as the timely application of evidence-based medical and surgical concepts designed to maintain a patient's hemoglobin (Hb) concentration, optimize hemostasis and minimize blood loss in an effort to improve the outcomes. More in detail, PBM focuses on three pillars:

* optimizing red cell mass;
* minimizing blood loss and bleeding;
* optimizing tolerance of anemia.

The implementation of the three pillars of PBM leads to improved patient' outcomes by relying on his/her own blood rather than on that of a donor. PBM goes beyond the concept of appropriate use of blood products, because it precedes and strongly reduces the use of transfusions by correcting modifiable risk factors long before a transfusion may even be considered. Importantly, the PBM is transversal to diseases, procedures and disciplines. It is solely aimed at managing a patient's resource (i.e., his/her blood), shifting the attention from the blood component to the patient himself/herself.

The recent and growing interest in PBM is principally driven by its notable impact on several outcomes. According to different studies PBM is able to reduce mortality up to 68%, reoperation up to 43%, readmissions up to 43%, composite morbidity up to 41%, infection rate up to 80%, average length of stay by 16 to 33%, transfusion from 10% to 95%, and costs from 10% to 84% (dependently from the healthcare system). Consistently, from patient's safety and better outcomes, the PBM achieves the aim of costs saving and fast-track policies adoption, satisfying some key performance indicators. In this sense, there clearly appears to be an extraordinary similitude between ERAS and PBM programs: they are both multidisciplinary and multifactorial, both centered on the patient, embracing the entire perioperative period, both evidence-based, both offering measurable positive influence on early outcomes after surgery. Actually, most recent guidelines on ERAS programs in colorectal surgery include preoperative anemia management in their suggested items. Finally, although the available evidence strongly suggests that the adoption of ERAS and PBM programs may lead to a significant improvement of outcomes, there still are no studies investigating the effects of adherence to the two programs. Therefore, the Italian ColoRectal Anastomotic Leakage (iCral) study group decided to design this prospective study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients submitted to laparoscopic/robotic/open/converted ileo-colo-rectal resection with anastomosis, including planned Hartmann's reversals.
2. American Society of Anesthesiologists' (ASA) class I, II, III or IV
3. Elective or delayed urgency (> 24 hours from admission) surgery
4. Patients' written acceptance to be included in the study.

Exclusion Criteria:

1. American Society of Anesthesiologists' (ASA) class V
2. Emergent surgery (≤ 24 hours from admission)
3. Pregnancy
4. Hyperthermic intraperitoneal chemotherapy for carcinomatosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing elective colorectal surgery with anastomosis will be included in a prospective database after written informed consent.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage rate | within 8 weeks from the operation
  number of patient with anastomotic leakage
Major morbidity rate | within 8 weeks from the operation
  number of patient with any Clavien-Dindo grade > II adverse event
Transfusion rate | from 4 weeks before to 8 weeks after the operation
  number of patient receiving at least one unit of packed red blood cells

SECONDARY OUTCOMES:
Overall morbidity rate | within 8 weeks from the operation
  number of patient with any adverse event
Length of Postoperative Hospital Stay (LOS) | within 8 weeks from the operation
  Total number of days spent in the hospital (including any readmission)
Number of transfused blood units | from 4 weeks before to 8 weeks after the operation
  Total number of transfused blood units
Postoperative hemoglobin values | 4 days after the operation, at discharge, 6 weeks after the operation
  Values of Hemoglobin (g/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Sandro Pertini, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No
Anonymized participant-level datasets will be available after study completion upon reasonable request by contacting the principal investigator.